CLINICAL TRIAL: NCT01266915
Title: Molecular Studies on Cutaneous Lupus
Brief Title: Cutaneous Lupus Registry
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ben Chong, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 112008-008
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Lupus Erythematosus
Keywords: SCLE; CLE; DLE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: Normal disease free (non lupus) subjects
- Diseased Control
- Diseased group 1: Those subjects with systemic lupus erythematosus.
- Diseased group 2: Subjects diagnosed with cutaneous lupus.

SUMMARY:
Approximately 1.4 million individuals in the United States have systemic lupus erythematosus, and about 85% of these individuals develop skin lesions at some point of their disease. Cutaneous lupus erythematosus represents the skin manifestations of systemic lupus erythematosus, and can appear in people with or without systemic lupus. It is a mentally, physically, and emotionally debilitating disease that affects both the quality of life and social well-being of those affected.

The cause of cutaneous lupus is not completely understood, but likely includes multiple factors from our genes and the environment. Multiple genetic studies with small numbers of cutaneous lupus patients have been performed to determine which genes are associated with cutaneous lupus. This study aims to accumulate even larger numbers of patients to confidently identify genes and the proteins they encode that could contribute greatly to the formation of cutaneous lupus. The discovery of these genes and proteins would help not only uncover how cutaneous lupus forms, but also improve our abilities to diagnose this disease and predict its course, and stimulate new drug development.

DETAILED DESCRIPTION:
The purpose of this study is to create a national registry of patients with cutaneous lupus patients in order to address many unknown questions about this disease. Specifically, we are interested in better understanding the causes of cutaneous lupus and improving our methods of diagnosis, prognosis, and management of this disease. We plan to use information from all patient sources, including medical histories, clinical information, laboratory data, and blood and skin samples in order to answer these questions.

Each study patient will be asked to complete a series of questionnaires, which, for example, will ask about cutaneous and/or systemic lupus history, past medical history, family history, quality of life, and sun protective habits. Patients will be also asked to donate blood and skin samples and undergo digital photography of affected areas. No treatments will be administered as part of this study, but all participants will be notified of clinical trials being conducted at UT Southwestern. This study is for the purpose of data collection only. Patients will be asked to be followed on an annual basis for five years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cutaneous lupus erythematosus and/or systemic lupus erythematosus by clinical, laboratory, and histopathological findings
* Ability to speak and read English or Spanish at a 6th grade reading level (a translator will be available with additional consent forms in Spanish)
* Ability to give written informed consent

Exclusion Criteria:

* Less than 18 years of age, since the characteristics of the disease in these subjects could be very different
* Due to a medication, in which its discontinuation results in the resolution of cutaneous lupus, since the characteristics of the disease in these subjects could be very different
* Medical conditions who do not warrant a skin biopsy
* Unable to give written, informed consent or undergo a skin biopsy and/or venipuncture for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with Lupus Erythematosus
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Genes | 5 years
Proteins (ie. signaling proteins, autoantibodies) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center Dallas, Dallas, Texas, United States